CLINICAL TRIAL: NCT06595758
Title: Effects of Pharmacogenetics on Pharmacokinetics and Toxicity of Doxorubicin in Egyptian Breast Cancer Patients
Brief Title: This Study Investigates the Impact of Single Nucleotide Polymorphisms in Genes Involved in the Pharmacokinetics and Toxicity of Doxorubicin (DOX) in Egyptian Female Patients with Breast Cancer. It Also Aims to Explore the Association of Pretreatment Neutrophil to Lymphocyte Ratio to PCR
Status: Completed | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Naglaa Fathy Mohamed Ebaid, Assistant Lecturer of clinical pharmacy, Menoufia University
Other Study IDs: Egyptian breast cancer patient
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: Doxorobicin; Pharmacokinetics; SLC22A16; CBR1; SNPs; Toxicity; Neoadjuvant chemotherapy; Pathological complete response; Neutrophil to lymphocyte ratio
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to investigate the effect of single nucleotide polymorphisms (SNPs) of genes involved in doxorubicin transport and metabolism on its pharmacokinetics and toxicity in Egyptian breast cancer patients.

It also aims to explore the association of pretreatment neutrophil to lymphocyte ratio (NLR) with pathological complete response (pCR).

DETAILED DESCRIPTION:
Plasma concentrations of doxorubicin will be determined and venous blood samples will be obtained from each patient for SNP genotyping of genes involved in doxorubicin transport and metabolism on its pharmacokinetics and toxicity in Egyptian breast cancer patients [prospective study].

A complete blood count was carried out at baseline for patients receiving neoadjuvant chemotherapy. The neutrophil to lymphocyte ratio (NLR) was calculated as the ratio between the absolute count of neutrophils and the absolute count of lymphocytes [ retrospective study].

ELIGIBILITY:
Inclusion Criteria:

* Females aged ≥ 18 years
* Performance status 0 or 1
* No contraindication to chemotherapy
* Adequate bone marrow
* Adequate hepatic function
* Adequate renal function

Exclusion Criteria:

* Poorly controlled diabetes mellitus
* Ischemic heart disease
* Uncontrolled hypertension
* Active infections
* Baseline ejection fraction < 50%
* Performance status ≥ 2
* Pregnancy Lactation, bilateral breast cancer, male patients, primary surgery, distant metastases, other malignancies, inflammations, hematological disorders, autoimmune diseases, and patients taking non-steroidal anti-inflammatory drugs (NSAIDs), steroidal and antibiotic therapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female Egyptian patients with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Doxorubicin plasma concentrations | baseline
  Plasma concentrations of doxorubicin will be determined using a suitable analytical method.
neutrophil to lymphocyte ratio | baseline
  The neutrophil to lymphocyte ratio (NLR) was calculated as the ratio between the absolute count of neutrophils and the absolute count of lymphocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- Menofia university, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No
Only up on reasonable request

REFERENCES:
- [Background] Lal S, Wong ZW, Jada SR, Xiang X, Chen Shu X, Ang PC, Figg WD, Lee EJ, Chowbay B. Novel SLC22A16 polymorphisms and influence on doxorubicin pharmacokinetics in Asian breast cancer patients. Pharmacogenomics. 2007 Jun;8(6):567-75. doi: 10.2217/14622416.8.6.567. PMID 17559346
- [Background] Speth PA, van Hoesel QG, Haanen C. Clinical pharmacokinetics of doxorubicin. Clin Pharmacokinet. 1988 Jul;15(1):15-31. doi: 10.2165/00003088-198815010-00002. PMID 3042244
- See also: Development of a predictive model utilizing the neutrophil to lymphocyte ratio to predict neoadjuvant chemotherapy efficacy in early breast cancer patients — https://pubmed.ncbi.nlm.nih.gov/33446717/